CLINICAL TRIAL: NCT02826941
Title: Moderate Hypothermia in Neonatal Hypoxic Ischemic Encephalopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Dorothea D. Jenkins, Associate Professor of Pediatrics, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NS38062; R01NS038062 (NIH)
Record Dates: First submitted 2016-05-23; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Neonatal Asphyxial Encephalopathy; Hypoxic Ischemic Encephalopathy
Keywords: hypothermia treatment
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia (Experimental): If randomized to hypothermia, plastic bags filled with ice wrapped in a washcloth were applied to the head and body for approximately 2 hours, then the infant was placed on an adult-size, water-circulating, cooling blanket (Cincinnati Sub-Zero Blanketrol II®, Cincinnati, OH), servo-controlled to rectal temperature to 33 ± 0.5 °C for 48 hours at the participating tertiary care center. Rewarming by 0.5°C per hour was begun after 48 hours of hypothermia.
  Interventions: Other: hypothermia
- Normothermia (Placebo Comparator): If randomized to normothermia, rectal temperatures were maintained at 37 ± 0.5 °C per standard neonatal intensive care unit practice, using adult-size, water-circulating, cooling blanket (Cincinnati Sub-Zero Blanketrol II®, Cincinnati, OH), servo-controlled to rectal temperature of 37 ± 0.5 if baby was febrile.
  Interventions: Other: normothermia

INTERVENTIONS:
Other: hypothermia — Systemic hypothermia by Cincinnati Sub-Zero Blanketrol II®, servo-controlled to 33.0 degrees C rectal temperature, started within 6hours of hypoxic ischemic birth, and continued for 48hours
  Other Names: whole body cooling
  Arms: Hypothermia
Other: normothermia — Rectal temperatures in neonates receiving normothermia were maintained at 37.0+or -0.5 degrees C, using overhead warmer or Cincinnati Sub-Zero Blanketrol II®, servo-controlled to rectal temperature of 37.0 degrees C.
  Arms: Normothermia

SUMMARY:
This study was a multicenter, randomized, controlled pilot trial of moderate systemic hypothermia (33°C) vs normothermia (37°C) for 48 hours in infants with neonatal encephalopathy instituted within 6 hours of birth or hypoxic-ischemic event.

DETAILED DESCRIPTION:
The trial tested the ability to initiate systemic hypothermia in outlying hospitals and participating tertiary care centers, and determined the incidence of adverse neurologic outcomes of death and developmental scores at 12 months by Bayley II or Vineland tests between normothermic and hypothermic groups. This trial identified potential safety outcomes, compared the adverse effects of hypothermia among hypoxic-ischemic encephalopathy (HIE) infants in the normothermic and hypothermic treatment groups, and obtained rates of adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

One clinical indication of hypoxic-ischemic injury

* cord gas pH ≤ 7.0 or base deficit ≥13,
* initial infant gas pH < 7.1,
* Apgar score ≤5 at 10 minutes,
* continued resuscitation after 5 min,
* fetal bradycardia with heart rate < 80 beats per minute lasting ≥15 min,
* postnatal event O2 sat <70% or arterial O2<35 for 20 min with ischemia

And two neurologic findings of neonatal encephalopathy, abnormalities of:

* tone,
* reflexes,
* state of consciousness,
* seizures,
* posturing,
* autonomic dysfunction

Exclusion Criteria:

* Maternal chorioamnionitis,
* sepsis at birth,
* birth weight or head circumference <10%,
* presumed chromosomal abnormality

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 1999-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Death or severely abnormal Psychomotor Development Index scores on Bayley II | 12 months
  Death or severe outcomes

SECONDARY OUTCOMES:
bradycardia | 0-96 hours
  number of patients with heart rate < 80 bpm

OTHER OUTCOMES:
coagulopathy | 1-4 days of life
  Mean Prothrombin time
Death | by 12 months of age
  numbers of patients who are withdrawn from support or die from multiorgan system failure

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea D Jenkins, MD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: Yes
upon request

REFERENCES:
- [Result] Eicher DJ, Wagner CL, Katikaneni LP, Hulsey TC, Bass WT, Kaufman DA, Horgan MJ, Languani S, Bhatia JJ, Givelichian LM, Sankaran K, Yager JY. Moderate hypothermia in neonatal encephalopathy: efficacy outcomes. Pediatr Neurol. 2005 Jan;32(1):11-7. doi: 10.1016/j.pediatrneurol.2004.06.014. PMID 15607598
- [Result] Eicher DJ, Wagner CL, Katikaneni LP, Hulsey TC, Bass WT, Kaufman DA, Horgan MJ, Languani S, Bhatia JJ, Givelichian LM, Sankaran K, Yager JY. Moderate hypothermia in neonatal encephalopathy: safety outcomes. Pediatr Neurol. 2005 Jan;32(1):18-24. doi: 10.1016/j.pediatrneurol.2004.06.015. PMID 15607599
- [Result] Jenkins DD, Lee T, Chiuzan C, Perkel JK, Rollins LG, Wagner CL, Katikaneni LP, Bass WT, Kaufman DA, Horgan MJ, Laungani S, Givelichian LM, Sankaran K, Yager JY, Martin R. Altered circulating leukocytes and their chemokines in a clinical trial of therapeutic hypothermia for neonatal hypoxic ischemic encephalopathy*. Pediatr Crit Care Med. 2013 Oct;14(8):786-95. doi: 10.1097/PCC.0b013e3182975cc9. PMID 23897243
- [Result] Jenkins DD, Rollins LG, Perkel JK, Wagner CL, Katikaneni LP, Bass WT, Kaufman DA, Horgan MJ, Languani S, Givelichian L, Sankaran K, Yager JY, Martin RH. Serum cytokines in a clinical trial of hypothermia for neonatal hypoxic-ischemic encephalopathy. J Cereb Blood Flow Metab. 2012 Oct;32(10):1888-96. doi: 10.1038/jcbfm.2012.83. Epub 2012 Jul 18. PMID 22805873